CLINICAL TRIAL: NCT02651610
Title: An Open-Label, Randomized, Phase II/III Trial of Taxane Therapy With or Without Bavituximab for the Treatment of HER2-Negative Metastatic Breast Cancer
Brief Title: Taxane Therapy With or Without Bavituximab for the Treatment of HER2-Negative Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 1401; 2015-003780-11 (EudraCT Number)
Record Dates: First submitted 2015-12-29; First posted 2016-01-11 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Breast Cancer
Keywords: PPHM 1401; bavituximab; Peregrine; Breast Cancer; HER-2 Negative; HER2 Negative
MeSH Terms: conditions — Breast Neoplasms | interventions — bavituximab; taxane; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taxane (Active Comparator): Docetaxel on Day 1 of 21-day cycles OR Paclitaxel on Days 1, 8, and 15 of 28-day cycles
  Interventions: Drug: Taxane
- Bavituximab plus taxane (Experimental): Bavituximab 3 mg/kg weekly PLUS Docetaxel on Day 1 of 21-day cycles OR Paclitaxel on Days 1, 8, and 15 of 28-day cycles
  Interventions: Biological: Bavituximab; Drug: Taxane

INTERVENTIONS:
Biological: Bavituximab — Biological: bavituximab
  Arms: Bavituximab plus taxane
Drug: Taxane — Drug: Taxane Other names: Paclitaxel. Taxotere, Taxotere, Docecad, Taxol
  Other Names: Paclitaxel; Taxotere; Docetaxel; Docecad; Taxol

SUMMARY:
The primary purpose of this research study is to see whether adding bavituximab (an investigational drug) to the standard chemotherapy drug taxane, will improve the results of the treatment for HER2-negative metastatic breast cancer.

DETAILED DESCRIPTION:
This is an open-label randomized trial in patients with HER2-negative metastatic breast cancer. Patients will be treated with either taxane alone (investigator choice of paclitaxel or docetaxel) or taxane with bavituximab. Paclitaxel will be given 3 of 4 weeks, docetaxel will be given once every 3 weeks, and bavituximab will be given weekly. All therapy will continue until disease progression, toxicity, withdrawal or consent, investigator decision, or study termination. Efficacy (overall response rate) is the primary endpoint while safety is the secondary endpoint.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent obtained prior to screening.
2. Females or males at least 18 years of age.
3. Histologically or cytologically documented metastatic HER2-negative breast cancer.
4. Measurable disease per RECIST 1.1 (Phase II); evaluable disease (Phase III)
5. ECOG performance status of 0 or 1.
6. Adequate hematologic function: absolute neutrophil count ≥1500 cells/µL; hemoglobin ≥9 g/dL; platelets ≥100,000/µL.
7. Adequate renal function: serum creatinine ≤1.8 mg/dL or calculated creatinine clearance >50 mL/min using the Cockcroft-Gault equation.
8. Adequate hepatic function: total bilirubin ≤ upper limit of normal (ULN), serum albumin ≥3.0 g/dL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5 × ULN. ALT and/or AST may be ≤5 × ULN if due to liver metastases. If ALT or AST is >1.5 and ≤5 × ULN in patients with liver metastases, alkaline phosphatase must be ≤2.5 × ULN. Patients with Gilbert's syndrome are allowed if total bilirubin is ≤2 × ULN and direct bilirubin is ≤ULN.
9. Prothrombin time (PT) and/or international normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) ≤1.5 × ULN if patient is not on anticoagulant therapy (a therapeutic PT and/or INR and aPTT is acceptable if the patient is on anticoagulants).
10. Patients must have a negative serum human chorionic gonadotropin test within 1 week of Day 1 (pregnancy test not required for patients with bilateral oophorectomy and/or hysterectomy or for those patients who are >1 year postmenopausal).
11. All patients of reproductive potential (ie, not surgically sterile or postmenopausal) must agree to use a highly effective method of contraception (<1% failure rate per year) during and 3 months after end of study treatment (female) or during and 6 months after the end of study treatment (male).

Exclusion Criteria

1. HER2-positive breast cancer.
2. Less than 6 months since last dose of prior adjuvant non-taxane regimen.
3. Less than 12 months since last dose of prior adjuvant taxane-containing regimen.
4. Any chemotherapy regimen for MBC within 3 weeks before Day 1.
5. Known history of bleeding diathesis or coagulopathy (eg, von Willebrand disease or hemophilia).
6. Bleeding:

   * Clinically significant bleeding, such as gross hematuria, gastrointestinal bleeding, and hemoptysis within the 6 months before screening, unless the cause has been identified and adequately treated (eg, cystitis, ulcer).
   * Minor biopsy-related bleeding lasting <24 hours and resolved at least 1 week before Day 1 is allowed.
7. Thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, arterial thrombosis) within 6 months before screening.
8. Grade 2 or higher peripheral neuropathy (eg, numbness, tingling, and/or pain in distal extremities).
9. Radiotherapy within 1 week preceding Day 1; ongoing acute toxicity from prior radiotherapy.
10. Either symptomatic or clinically active brain metastases (ie, requiring ongoing treatment). Patients are eligible if brain metastases are adequately treated. Patients must be either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent).
11. Major surgery within 4 weeks of Day 1.
12. Uncontrolled intercurrent disease (eg, diabetes, hypertension, thyroid disease, active infections).
13. Autoimmune disease, being treated with immunosuppressive drugs (eg, methotrexate or biological agents), or other conditions requiring immunosuppressive therapy (eg, prior allotransplantation).
14. History of hypersensitivity to bavituximab, docetaxel, paclitaxel, or to any of their excipients.
15. Symptomatic coronary artery disease, cerebrovascular accident or transient ischemic attack, myocardial infarction, arterial embolism, or unstable angina pectoris within 6 months of screening.
16. Currently pregnant, nursing, or planning a pregnancy during the study.
17. Investigational therapy within 28 days prior to Day 1.
18. Patient has a condition or is in a situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 24 months

SECONDARY OUTCOMES:
Safety Measures - Adverse Events and Laboratory Evaluations | 24 months
Efficacy: Disease Control Rate (DCR) | 24 Months
Efficacy: Duration of Response (DOR) | 24 Months
Efficacy: Progression Free Survival (PFS) | 24 Months
Efficacy: Overall Survival | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Study Chair — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Peregrine Pharmaceuticals Investigational Site, Bakersfield, California
  - Peregrine Pharmaceuticals Investigational Site, Tinley Park, Illinois